CLINICAL TRIAL: NCT06518317
Title: Short Versus Long Antiplatelet Therapy After TAVI
Acronym: SOLOTAVI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-508208-40-00
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Transcatheter Aortic Valve Replacement
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, blinded endpoint assessment, randomized non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: Multicenter, open label, blinded endpoint assessment, randomized non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short treatment (Experimental): Single antiplatelet therapy 75 to 100 mg aspirin for 3 months after TAVI followed by aspirin discontinuation
  Interventions: Drug: Aspirin
- long treatment (Active Comparator): Long term (lifetime) single antiplatelet therapy75 to 100 mg aspirin therapy after TAV
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Short duration of aspirin (3 months) is compared to long duration of aspirin (12 months)

SUMMARY:
The goal of this clinical trial is to learn if reducing the duration of treatment by aspirin to 3 months (short treatment regimen) after percutaneous aortic valve replacement is as safe and efficient as the routine lifetime treatment by aspirin (standard treatment regimen).

The main questions it aims to answer are:

Does the reduction of the duration of aspirin reduces rates of bleeding without increasing the risk of cardiovascular events.

Researchers will compare a short treatment by aspirin (3 months) to a long treatment by aspirin (12 months) after percutaneous replacement of the aortic valve.

Participants will:

Take aspirin for 3 months in one group or 12 months in another group Be contacted by phone or visit the clinic at 3, 4, 6, 8, 10 and 12 months after hospital discharge Keep a diary of any bleeding or cardiovascular events occurring during the study period

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Aortic stenosis (AS) is the most common heart valve disease requiring intervention among elderly patients. Surgical aortic valve replacement which was the only curative treatment of AS has been challenged during the past decade by the trans-aortic valve implantation (TAVI) which is becoming the first line treatment of such condition.

Antithrombotic therapy after TAVI remains a matter of debate. In patients with no indication for antiplatelet therapy, aspirin alone is recommended for lifetime. However, after bioprosthetic surgical valve replacement, aspirin is to be discontinued 3 months after surgery and there is no evidence that it should be continued in patients after TAVI with no other indication for such therapy (more than half of low risk and a third of intermediate risk TAVI patients). Aspirin as compared to placebo in the setting of primary prevention is associated with a 38% relative risk increase of major bleeding in elderly patients with no benefit in terms of mortality or cardiovascular events.

Hence there is a major gap of knowledge on whether aspirin is beneficial or harmful if continued more than 3 months as recommended after successful TAVI in absence of another indication, as most such patients are elderly and at high bleeding risk.

STUDY POPULATION Adult patients with successful transfemoral TAVI for symptomatic aortic stenosis with no indication for long term antiplatelet or anticoagulant therapy. This represents approximately 30% of the TAVI patient population.

STUDY DESIGN Multicenter, open label, blinded endpoint assessment, randomized non-inferiority trial nested in an ongoing prospective nationwide registry RANDOMIZATION All potentially eligible patients will be included after successful TAVI at hospital discharge to be randomized to receive the experimental or control strategy. Randomization will be performed at hospital discharge (visit 0) after revision of inclusion/exclusion criteria. Randomization will be stratified by center and type of valve (balloon expandable or self-expandable). A hierarchical test procedure will be used for the analysis of the endpoints. A hierarchical test procedure will be used for the analysis of the primary and principal secondary endpoints.

EXPERIMENTAL ARM Single antiplatelet therapy 75 to 100 mg aspirin for 3 months after TAVI followed by aspirin discontinuation CONTROL ARM Long term (lifetime) single antiplatelet therapy75 to 100 mg aspirin therapy after TAVI PRIMARY END POINT Net clinical benefit defined by the composite of all cause death, myocardial infarction, ischemic or hemorrhagic stroke and major or disabling bleeding assessed at 12 months follow-up NUMBER OF PATIENTS TO BE INCLUDED 1400 (700 in each group)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Male or, post-menopausal -with no menses for 12 months without an alternative medical cause- or permanently sterilized -hystercetomy, bilateral salpingectomy or bilateral oophorectomy- female
* Successful transfemoral TAVI for symptomatic aortic stenosis as defined by VARC-33

  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device (excluding permanent pacemaker) or to a major vascular or access-related, or cardiac structural complication
* Written informed consent
* Social security affiliated
* French speaking

Exclusion Criteria:

* Un-successful TAVI defined by the absence of any of the above-mentioned criteria defining successful TAVI3
* Alternative non-femoral-approach TAVI: apical, direct trans-aortic, subclavian, axillary or carotid approaches
* TAVI for other indications than aortic stenosis (pure aortic regurgitation)
* Valve in valve TAVI
* Any indication for long term antiplatelet therapy: (e.g. coronary artery disease, cerebrovascular disease, peripheral arterial disease…) at any time prior to randomization
* Any indication for oral anticoagulation: (e.g. atrial fibrillation, deep vein thrombosis, pulmonary embolism, ventricular thrombus…) at any time prior to randomization
* Patients on long term antiplatelet or anticoagulant therapy prior to TAVI for any other indication than TAVI
* Any contraindication to long term antiplatelet therapy (e.g. allergy or intolerance to aspirin, major bleeding, high bleeding risk, thrombocytopenia < 50 000, major haemostasis disorder…)
* Women of childbearing potential: non menopaused -with no menses for 12 months without an alternative medical cause- and not permanently sterilized -hystercetomy, bilateral salpingectomy or bilateral oophorectomy-
* Adult with protective measures (tutorship, curatorship)
* Patients considered as vulnerable by the investigators because of medical, psychological or social conditions:

  * Patients with known or discovered severe cognitive impairment
  * Patients with treated or untreated severe psychological or psychiatric conditions
  * Patients with uncorrected severe hearing or visual handicap
  * Patients with addictive alcohol, drug or substance abuse
  * Patients with protective measures (guardianship, tutorship, curatorship)
  * Any other condition considered by the investigators as not warranting informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Net clinical benefit | 12 months after randomisation
  The composite of all cause death, type 1 myocardial infarction, NeuroARC types 1a, 1aH, 1b, 1c, 1d ischemic or hemorrhagic central nervous system injury and non-procedure-related major or disabling bleeding VARC 3 types 2 or 3

SECONDARY OUTCOMES:
Non-procedure-related bleeding | 12 months
  VARC 3 classification 1 to 4 bleeding
Major or disabling or life threatening bleeding | 12 months
  VARC 3 classification 2 or 3 bleeding
Major cardiovascular events | 12 months
  The composite of all cause death, type 1 myocardial infarction based on the universal definition or stroke defined by NeuroARC types 1a, or 1d ischemic CNS injury

OTHER OUTCOMES:
Minor bleeding | 12 months
  Type 1 VARC 3 classification bleeding
Major bleeding | 12 months
  Type 2 VARC 3 classification bleeding
Disabling or life threatening bleeding | 12 months
  Type 3 VARC 3 classification bleeding
Fatal bleeding | 12 months
  Type 4 VARC 3 classification bleeding
Death | 12 months
  Death of any cause
Cardiovascular death | 12 months
  Death of cardiovascular cause
Myocardial infarction | 12 months
  Type 1 myocardial infarction based on the universal definition
Ischemic Stroke | 12 months
  NeuroARC types 1a, or 1d ischemic CNS injury
Intracranial bleeding | 12 months
  NeuroARC type 1aH, 1b, 1c hemorrhagic CNS injury
Transient cerebral ischemic attack | 12 months
  NeuroARC type 3a
Hospitalization | 12 months
  Hospitalization for any cause
Cardiovascular hospitalization | 12 months
  Hospitalization for cardiovascular causes as defined by VARC 3
clinically significant prosthetic valve thrombosis | 12 months
  VARC 3 classification -defined
Death at 2 years | 24 months
  Death assessed using the national mortality database

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
IPD sharing may be considered if authorised by PI and promoter